CLINICAL TRIAL: NCT03942510
Title: Autonomical and Hemodynamic Repercussions on Excentric Resistance in Different Intensities Associated With Blood Flow Restriction: a Randomized Clinical Trial
Brief Title: Autonomical and Hemodynamic Repercussions on Excentric Resistance in Different Intensities With Blood Flow Restriction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paulista University (Other)
Responsible Party: Principal Investigator, Franciele Marques Vanderle, Principal Investigator, Paulista University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: U1111-1232-0808
Record Dates: First submitted 2019-04-30; First posted 2019-05-08 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Exercise
Keywords: resistance training; vascular occlusion; hemodynamics, cardiovascular system; autonomic nervous system; heart rate; recovery of physiological function
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High intensity eccentric training (Experimental): high intensity (80% isometric peak) eccentric training of the knee extensors in the isokinetic will be performed during 6 weeks, 3 times a week.
  Interventions: Other: eccentric exercise with blood flow restriction
- High intensity eccentric training with blood flow restriction (Experimental): high intensity (80% isometric peak) eccentric training of the knee extensors in the isokinetic associated with a pressure cuff placed in the proximal thigh (40% of absolute occlusion pressure) will be performed during 6 weeks, 3 times a week.
  Interventions: Other: eccentric exercise with blood flow restriction
- Low intensity eccentric training (Experimental): A low intensity (40% isometric peak) eccentric training of the knee extensors in the isokinetic will be performed during 6 weeks, 3 times a week.
  Interventions: Other: eccentric exercise with blood flow restriction
- Low intensity eccentric training with blood flow restriction (Experimental): A low intensity (40% isometric peak) eccentric training of the knee extensors in the isokinetic associated with a pressure cuff placed in the proximal thigh (40% of absolute occlusion pressure)will be performed during 6 weeks, 3 times a week.
  Interventions: Other: eccentric exercise with blood flow restriction

INTERVENTIONS:
Other: eccentric exercise with blood flow restriction — High/low intensity eccentric training group (80% and 40% of isometric peak torque) with or not blood flow restriction.

SUMMARY:
Introduction: Studies on resistance training (RT) associated with blood flow restriction (BFR) have emerged as an alternative method of gaining strength and hypertrophy; however, the cardiovascular and autonomic repercussion of BFR at different intensities is unknown. Thus, it becomes relevant to investigate this type of training in post-exercise. Objective: investigate and compare autonomic and hemodynamic responses of acute eccentric RT with different intensities associated or not to BFR in healthy youngsters. Method: This is a randomized clinical trial including 60 healthy men aged 18-35 years, divided into four groups according to exercise intensity and BFR: 80% without BFR, 40% without BFR, 80% with BFR and 40% with BFR. Exercise intensity will be determined by the peak of excentric torque on the dinamometer isokinetic method and by the BFR, as being 40% of the intensity required for the complete examination of the blood flow evaluated by Doppler. Participants will do an eccentric femoral quadriceps muscle exercise session on the isokinetic dynamometer according to the previously randomized group. For recovery analyzes, the recovery heart rate (HRR) in the 1st (HRR1) and 2nd (HRR2) minute, rMSSD of 30 seconds, the hemodynamic parameters (heart rate, systolic and diastolic blood pressure, respiratory rate, peripheral oxygen saturation and rate pressure product) and heart rate variability (HRV) indices analyzed in the time domain (mean HR, rMSSD and SDNN), frequency domain (LF and HF [nu and ms2]) and Poincaré plot (SD1 and SD2). The analysis will be occur on baseline, immediately e after the excentric exercise and in the post exercise period for 60 minutes. Descriptive statistics method and comparison of HRV indices and hemodynamic parameters between moments and groups will be performed with the aid of the analysis of variance technique for the repetitive measures model without the schema of two sets of tests to follow . The level of significance will be p <0.05.

ELIGIBILITY:
Inclusion Criteria:

* male sex;
* healthy;
* aged between 18 and 35 years

Exclusion Criteria:

* smokers;
* alcoholics;
* use drugs that influenced cardiac autonomic activity;
* cardiovascular, metabolic or endocrine diseases.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2019-10-17 (Actual); Study Completion 2020-12-22 (Actual)

PRIMARY OUTCOMES:
heart rate variability indices in the time domain | Change from baseline at 3rd week and 6rd week
  mean HR, rMSSD and SDNN in ms
heart rate variability indices analyzed in the Poincaré plot | Change from baseline at 3rd week and 6rd week
  SD1 and SD2 in ms
heart rate variability indices in the frequency domain | Change from baseline at 3rd week and 6rd week
  LF and HF in nu and ms2
vagal reentry | Change from 1 day at 10 day and 18 day
  rMSSD of 30 seconds in ms
heart rate recovery | Change from 1 day at 10 day and 18 day
  the recovery heart rate (HRR) in the 1st (HRR1) and 2st (HRR2) minute [bpm]

SECONDARY OUTCOMES:
hemodynamic parameter | through study completion, an average of 6 weeks
  heart rate [bpm]
hemodynamic parameter | through study completion, an average of 6 weeks
  systolic and diastolic blood pressure [mmHg]
hemodynamic parameter | through study completion, an average of 6 weeks
  respiratory rate [irpm]
hemodynamic parameter | through study completion, an average of 6 weeks
  peripheral oxygen saturation [%]

CONTACTS AND LOCATIONS:
Overall Officials: Franciele M Vanderlei, PhD, Principal Investigator — Paulista State University
Locations (1):
- Leonardo Kesrouani Lemos, Presidente Prudente, São Paulo, Brazil